CLINICAL TRIAL: NCT03029078
Title: FEcal Transplant, a Hope to Eradicate Colonization of Patient Harboring eXtreme Drug Resistant Bacteria?
Acronym: FEDEX
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centre d'Investigation Clinique et Technologique 805 (Other)
Responsible Party: Principal Investigator, Benjamin DAVIDO, M.D, M.S, Centre d'Investigation Clinique et Technologique 805
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GIPIT002; 2014-003048-11 (EudraCT Number)
Record Dates: First submitted 2017-01-20; First posted 2017-01-24 (Estimated); Last update posted 2021-07-27 (Actual); Status verified 2021-07

CONDITIONS: Microbial Colonization; Bacterial Peritonitis; Faeces Smearing
Keywords: XDR; fecal microbiota transplant; eradicate; colonization; CRE; GRE; bacteria
MeSH Terms: conditions — Communicable Diseases | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Intervention Model Description: Pilot study of patients colonized by either CRE or GRE will be enrolled in order to evaluate the impact of fecal microbiota transplant on the eradication of XDR bacteria colonization
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fecal transplantation (Experimental): Patient will be transplanted with a healthy donor microbiota, free from XDR bacteria, in order to evaluate the impact on the digestive tract colonization Whole process of feces screening and reconstitution was under the responsibility of the pharmacists in charge of the study.
  Patient will benefit of a naso-duodenal tube in order to perform a bowel lavage prio to the fecal microbiota transplant.
  Patient will be monitored for 24h to rule out potential adverse events.
  Interventions: Drug: fecal microbiota transplant

INTERVENTIONS:
Drug: fecal microbiota transplant — We will perform a fecal microbiota transplant for patients harboring XDR bacteria in their digestive tract
  Other Names: FEDEX

SUMMARY:
Our trial try to eradicate digestive tract colonization of patient harboring Extreme Drug Resistant (XDR) bacteria by performing a fecal transplantation.

DETAILED DESCRIPTION:
Main objective:

Evaluate the eradication of the colonization of patient harboring XDR bacteria after a fecal transplantation from a healthy donor.

Secondary objectives:

English Evaluate the side effects of this procedure and tolerability. Evaluate the efficacy of the transplant if the patient is harboring glycopeptid resistant enteroccus (GRE) or carbapenem resistant enterobacteriae (CRE)

ELIGIBILITY:
Inclusion Criteria:

* Patient harboring a VRE or CRE bacteria
* Colonization confirmed by our microbiology department, including at least 3 positives swabs in the last month

Exclusion Criteria:

* Pregnant woman or breastfeeding
* immunosuppression including AIDS, corticosteroids over 60mg/day
* ongoing antibiotic treatment at the day of inclusion
* impossibility to obtain a signed consent form.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2014-11-01 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
Negativation of digestive tract colonization | At one week, 2 weeks, one month up to 6 months
  Negativation of the rectal swab performed, free from CRE or GRE

SECONDARY OUTCOMES:
Metagenomics profile between donor and recipient depending on decolonization | At one week, 2 weeks, one month up to 3 months
  Study with a universal super donor in order to improve efficacy

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Davido, MD, MS, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hopital Raymond Poincaré, Garches, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- Available data/document: Study Protocol — https://www.clinicaltrialsregister.eu/ctr-search/trial/2014-003048-11/FR